CLINICAL TRIAL: NCT02172274
Title: A Phase I, Open-label, Single-dose Trial to Investigate the Metabolism and Pharmacokinetics of 50 mg [14C]-BI 10773 When Administered as Oral Solution to Healthy Male Volunteers
Brief Title: BI 10773 Administered as Oral Solution to Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1245.8
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (1):
- [14C]-BI 10773 - oral solution (Experimental)
  Interventions: Drug: [14C]-BI 10773 - oral solution

INTERVENTIONS:
Drug: [14C]-BI 10773 - oral solution

SUMMARY:
Study to determine the pharmacokinetics of BI 10773 and total radioactivity including excretion mass balance, excretion pathways and metabolism following the oral administration of [14C] BI 10773

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to a complete medical history, including a physical examination, vital signs (blood pressure, pulse rate), 12-lead ECG (electrocardiogram), and clinical laboratory tests
* Age 18 to 55 years, inclusive
* Body mass index 18.5 to 29.9 kg/m2, inclusive
* Nonsmoker
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* Any finding in the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, hormonal, psychiatric or neurological disorders (including all forms of epilepsy)
* Surgery of the gastrointestinal tract (except appendectomy)
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Subjects with Gilbert's Syndrome
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within one month prior to administration of the trial drug
* Use of prescription medication, over-the-counter drugs or herbal preparations within 14 days prior to administration of the trial drug
* Participation in another trial with an investigational drug within two months prior to administration of the trial drug or during the trial
* History or evidence of habitual tobacco or nicotine use within six months prior to administration of the trial drug
* Alcohol abuse (more than 60 g/day)
* Drug abuse in opinion of investigator
* Blood donation (more than 100 mL within four weeks prior to administration of trial drug or during the trial)
* Excessive physical activity within five days prior to administration of trial drug
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial centre
* A marked baseline prolongation of QT/QTc interval (corrected QT interval)(e.g., repeated demonstration of a QTc interval >450 ms)
* Male subjects must agree to minimise the risk of female partners becoming pregnant from the dosing day until three months after the completion of the study. Acceptable methods of contraception for male volunteers include a vasectomy no less than three months prior to dosing, barrier contraception, or a medically accepted contraceptive method. For female partners of male volunteers, acceptable methods of contraception include intrauterine device, tubal ligation, hormonal contraceptive for at least two months, or diaphragm with spermicide
* Participation in more than one other radiolabeled investigational drug trial within one year prior to administration of the trial drug. The previous radiolabeled trial drug must have been received more than six months prior to administration of the trial drug for this study, and the total exposure from this study and the previous study will be within the recommended levels considered safe, per 21 CFR (Code of Federal Regulations) 361.1 (eg, less than 5000 mrem whole body annual exposure)
* Irregular defecation pattern (less than one bowel movement a day)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | pre-dose and up to 144 hours after administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | pre-dose and up to 144 hours after administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | pre-dose and up to 144 hours after administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to infinity) | pre-dose and up to 144 hours after administration
λz (terminal rate constant in plasma) | pre-dose and up to 144 hours after administration
t1/2 (terminal half-life of the analyte(s) in plasma) | pre-dose and up to 144 hours after administration
MRTpo (mean residence time of the analyte(s) in the body after oral administration) | pre-dose and up to 144 hours after administration
CL/F (apparent/total clearance of the analyte(s) in plasma after an extravascular dose) | pre-dose and up to 144 hours after administration
Vz/F (apparent volume of distribution during the terminal phase λz after an extravascular dose) | pre-dose and up to 144 hours after administration
feurine,0-tz (amount of analyte excreted in urine over the time interval from 0 to the time of the last quantifiable data point in % of dose, additionally excretion within each sampling interval will be calculated) | pre-dose and up to 168 hours after administration
fefaeces,0-tz (amount of analyte excreted in faeces over the time interval from 0 to the time of the last quantifiable data point in % of dose, additionally excretion within each sampling interval will be calculated) | pre-dose and up to 168 hours after administration
CLR,0-tz (renal clearance of analyte) | pre-dose and up to 168 hours after administration
Individual concentration-time profiles of [14C] radioactivity in whole blood, plasma, urine, and faeces | up to 8 days
Individual concentration-time profiles of BI 10773 in plasma and urine | up to 8 days
Rate and extent of excretion mass balance based on the total radioactivity in urine and faeces | up to 8 days
Identification of major metabolites in urine, faeces, and plasma | up to 8 days
Cblood cell/Cplasma ratio of [14C]-radioactivity | up to 8 days
Measurement of the plasma protein binding of total [14C] radioactivity in human plasma samples ex vivo | up to 8 days

SECONDARY OUTCOMES:
Number of patients with abnormal findings in physical examination | Baseline and within 6 days after discharge
Number of patients with clinically significant changes in vital signs (blood pressure, pulse rate) | Baseline, days 1, 2, 7 and within 6 days after discharge
Number of patients with abnormal findings in 12-lead electrocardiogram (ECG) | Baseline, days 1, 2, 7 and within 6 days after discharge
Number of patients with abnormal changes in laboratory parameters | Baseline, days 1, 2 and within 6 days after discharge
Number of patients with adverse events | Up to 22 days
Assessment of tolerability by investigator on a 4-point scale | Day 8